CLINICAL TRIAL: NCT02673268
Title: Robot Assisted Mastectomy Via Axillary Way With Areola Conservation and Immediate Reconstruction
Acronym: MARCI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-A00745-44; 2015/2250 (Other: CSET number)
Record Dates: First submitted 2016-02-01; First posted 2016-02-03 (Estimated); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Mastectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with breast cancer (Experimental)
  Interventions: Procedure: Mastectomy; Device: Da Vinci Robot Xi

INTERVENTIONS:
Procedure: Mastectomy
Device: Da Vinci Robot Xi

SUMMARY:
The objective of this study is to demonstrate the feasibility of a mastectomy with conservation of the areola using axillary way only with the Da Vinci Robot Xi and immediate breast reconstruction using prosthesis.

The interest is to avoid scars on the breast. The scars are limited to the armpit and under the arm.

The aim is also to study the rate of complications, cosmetic results and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1 .Patients with an indication of mastectomy with areola conservation 2. In case of carcinologic surgery:

* Disease located more than 2cm of the areola on the clinical and paraclinical evaluation
* Patients with indication of total mastectomy
* Patients looking for immediate reconstruction 3. In case of prophylactic surgery
* Patients wishing a prophylactic surgery because of highly risked mutation (BRCA1, BRCA2....) 4. Cup A, B or C maximum 5. Aged between 18 and 70 years old 6. OMS 0, 1 7. Signed informed consent 8. Patients affiliated to a social security system

Exclusion Criteria:

1. Patients with a high risk of skin necrosis
2. Planned post operative radiotherapy
3. Patients with an historic of breast surgery on the side that needs to be operated
4. Pregnant or breastfeeding women
5. Persons deprived of liberty
6. Persons not able to undergo medical follow up due to geographical, social or psychic reasons

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-11-25 (Actual); Primary Completion 2019-11 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Rate of necrosis | Assessed up to 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Gustave Roussy Cancer Campus, Villejuif, Val de Marne, France

REFERENCES:
- [Derived] Sarfati B, Struk S, Leymarie N, Honart JF, Alkhashnam H, Tran de Fremicourt K, Conversano A, Rimareix F, Simon M, Michiels S, Kolb F. Robotic Prophylactic Nipple-Sparing Mastectomy with Immediate Prosthetic Breast Reconstruction: A Prospective Study. Ann Surg Oncol. 2018 Sep;25(9):2579-2586. doi: 10.1245/s10434-018-6555-x. Epub 2018 Jun 29. PMID 29959612